CLINICAL TRIAL: NCT04685980
Title: Factors Associated With Failed Spinal Anesthesia for Cesarean Delivery, a Retrospective Case-control Study
Brief Title: Factors Associated With Failed Spinal Anesthesia for Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 290/2563 (EC1); 445/2020 (Other: Siriraj Institutional Review Board)
Record Dates: First submitted 2020-12-14; First posted 2020-12-28 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Adverse Effect; Cesarean Section Complications
Keywords: Spinal anaesthesia; cesarean section
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Failed spinal anaesthesia group: Failed spinal anaesthesia: failure of anaesthetic level of blockade both sensory and motor blockage, and consequently receive general anaesthesia
  Interventions: Procedure: spinal anaesthesia with local anaesthetic and intrathecal morphine
- Control Group: Patient receiving spinal anaesthesia and successfully finish the cesarean section
  Interventions: Procedure: spinal anaesthesia with local anaesthetic and intrathecal morphine

INTERVENTIONS:
Procedure: spinal anaesthesia with local anaesthetic and intrathecal morphine — Patients undergoing cesarean delivery and received spinal anaesthesia with local anaesthetic and intrathecal morphine

SUMMARY:
The aim of this study is to reveal the factor associated with failed spinal anaesthesia in cesarean delivery. We conduct the retrospective case-control study to elucidate the involving factors.

DETAILED DESCRIPTION:
Spinal anaesthesia is the anaesthetic technique of choice of patients undergoing cesarean delivery due to its rapid onset, good reliability and good efficacy. However, the inadequate or failed spinal anaesthesia can occur. The previous literatures revealed incidence of failed spinal anaesthesia was as high as 0.5-6%. Failure of spinal anaesthesia leads to numerous maternal and neonatal consequences. Those failed spinal anaesthesia patients required general anaesthesia with endotracheal tube which may cause several complications such as hypoxia, difficult intubation, failed intubation and pulmonary aspiration. Also, a recent network meta-analysis showed general anaesthesia decreasing neonatal Apgar score.

The factors that associated with failed spinal anaesthesia in cesarean delivery has been studied. The amount of local anaesthetic, needle type, patients' body mass index (obesity), and experiences of the anaesthetist performing spinal block influenced the failure of spinal anaesthesia. The details and factors of failed spinal anaesthesia in our hospital was scarce. It has not yet been published in the literature.

Therefore, the aim of this study is to reveal the factor associated with failed spinal anaesthesia in cesarean delivery. We conduct the retrospective case-control study to elucidate the involving factors.

ELIGIBILITY:
Inclusion Criteria:

* Age >,= 18 years
* Undergoing cesarean delivery
* Failed spinal anaesthesia and received general anaesthesia with endotracheal tube

Exclusion Criteria:

* Gestational age < 24 weeks
* Received combined spinal-epidural anaesthesia
* Received peripheral nerve blockade

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who gestational age > 24 weeks and patient age more than or equal to 18 years, undergoing cesarean delivery and received spinal anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Age | At starting operation
  Factors involving failed spinal anaesthesia for cesarean delivery: patient age
Body mass index | At starting operation
  Factors involving failed spinal anaesthesia for cesarean delivery: patient body mass index (BMI) : weight and height will be combined to report BMI in kg/m^2
Anaesthesiologist performing spinal anaesthesia | At starting anaesthesia
  Factors involving failed spinal anaesthesia for cesarean delivery: Anaesthesiologist performing spinal anaesthesia (resident or consultant)
Time starting of operation | At starting operation
  Factors involving failed spinal anaesthesia for cesarean delivery: at which time cesarean delivery starting to performed eg. in office hour or out of office hour

SECONDARY OUTCOMES:
Incidence of failed spinal anaesthesia for cesarean delivery | At starting operation
  Incidence of failed spinal anaesthesia for cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University, THAILAND
Locations (1):
- Anesthesiology department, Siriraj hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The plan to make individual participant data (IPD) available to other researchers was undecided

REFERENCES:
- [Result] Punchuklang W, Nivatpumin P, Jintadawong T. Total failure of spinal anesthesia for cesarean delivery, associated factors, and outcomes: A retrospective case-control study. Medicine (Baltimore). 2022 Jul 8;101(27):e29813. doi: 10.1097/MD.0000000000029813. PMID 35801788